CLINICAL TRIAL: NCT04227158
Title: The Association Between the Distributions MCH and RBC, and Mortality in a Cohort of Chronic Hemodialysis Patients: a 3-year Retrospective Observational Study
Brief Title: The Association Between the Distributions MCH and RBC, and Mortality in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Hyogo (Other)
Responsible Party: Principal Investigator, Yoshihiro Tsuji, visiting researche, Yoshihiro Tsuji, University of Hyogo
Other Study IDs: Uhyogo4
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-03

CONDITIONS: Renal Anemia
Keywords: red blood cell; mean corpuscular hemoglobin; hemoglobin; Hemodialysis patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients were classified into two groups based on the values of MCH and RBC, patients with MCH ≥30 pg but <35 pg and RBC ≤350×104/μL; and MCH <30 pg and RBC >350×104/μL. Associations between all-cause mortality and the distributions of MCH and RBC were assessed by Kaplan-Meier curves and Cox proportional hazards regression model.

DETAILED DESCRIPTION:
The Hb levels generally provides the value of RBC and iron status because mean corpuscular hemoglobin MCH is derived from the Hb divided by RBC. MCH depends on the size and concentration of erythrocytes. Thus, the value of RBC and MCH depend on dose of ESA and iron, respectively. Guidelines for Renal Anemia in Chronic Kidney Disease of 2015 Japanese Society for Dialysis Therapy recommend administration hemoglobin (Hb) levels ≥10 g/dL but <12 g/dL in dialysis patients.Patients whose Hb levels is maintained at 10 to 12 g/dL, Hb levels is widely distributed when divided into RBC and MCH. Therefore, the investigators examined the prognosis of life in the distribution of MCH and RBC.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be controlled with hemoglobin levels between ≥10 g/dL and <12 g/dL and had undergone maintenance HD for >1 year.

Exclusion Criteria:

* Patients will be excluded if they have peritoneal dialysis combined with HD, do not have records of laboratory investigations during this period, or are transferred to another hospital or lost to follow-up.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients has undergone maintenance Hemodialysis for >1 year.
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Survival rate between high or low RBC group (all cause death) | three years (retrospectively)
  Survival curves for 3-year survival, based on all available follow-up data, will perform with the use of Kaplan-Meier estimates and will be compared between groups with the use of the log-rank test, and used Holm's method as post hoc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuko MIZUNO, Ph.D., Study Director — University of Hyogo
Locations (1):
- Graduate School of Applied Informatics, University of Hyogo, Kobe, Hyōgo, Japan